CLINICAL TRIAL: NCT06713980
Title: Study on the Effects of Acupuncture on Pain, Acupoint Surface Temperature, and Meridian Energy Values in Patients with Cyclic Mastalgia
Brief Title: Study on the Effects of Acupuncture in Patients with Cyclic Mastalgia
Acronym: CM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuan Yu (Other)
Responsible Party: Sponsor-Investigator, Chuan Yu, Dr., Pinggu Hospital of Beijing Traditional Chinese Medicine Hospital
Organization: Pinggu Hospital of Beijing Traditional Chinese Medicine Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024pgzyy01; 2024pgzyy01 (Other Grant/Funding Number: Beijing Hospital)
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Breast Pain
MeSH Terms: conditions — Mastodynia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sham acupuncture group (Sham Comparator): In the SA group, non-penetrating sham acupuncture was applied at 14 specific non-acupuncture points on the back. A pedestal was affixed to each non-acupuncture point. Blunt-tip needles were then inserted into the pedestal at a depth of 3-5 mm, and it was ensured that they only touched the skin without penetration
  Interventions: Other: sham acupuncture
- acupuncture group (Experimental): the choice of acupoints was based on the theory of traditional Chinese medicine (TCM), as follows: Ashi point, Tanzhong (CV17), bilateral Wuyi (ST15), Rugen (ST18), Tianzong (SI11), Geshu (BL17), Ganshu (BL18), Hegu (LI4), Sanyinjiao (SP6), and Taichong (LR3).
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: sham acupuncture — In the sham acupuncture group, sham acupuncture was applied at 14 specific non-acupuncture points on the back.
  Arms: sham acupuncture group
Other: acupuncture — acupuncture:the choice of acupoints was based on the theory of traditional Chinese medicine (TCM). All needles were manually manipulated to achieve the deqi sensation
  Arms: acupuncture group

SUMMARY:
This study is designed to evaluate the effectiveness of acupuncture in treating cyclic mastalgia (breast pain that occurs in a cyclical pattern, often related to the menstrual cycle). The study will take place at the Pinggu District Traditional Chinese Medicine Hospital in Beijing and also included volunteers who are interested in participating. Sixty-six patients who meet the criteria for cyclic mastalgia will be chosen to take part in the study.The patients will be randomly divided into two groups: Observation Group (Acupuncture Group): 33 patients receive real acupuncture treatments.

Control Group (Sham Acupuncture Group): 33 patients receive sham acupuncture treatments.

This means that neither the participants nor the researchers know who is receiving the real or fake treatment, ensuring a fair comparison.

The study will last for 16 weeks. The main thing researchers look at is the change in daily average overall breast pain. Researchers also observe changes in:Infrared temperature at specific acupoints (Danzhong CV17, Rugen ST18, and Tianzong SI11).Meridian energy values of the Liver, Spleen, and Stomach meridians, which are concepts in Traditional Chinese Medicine related to the flow of energy in the body.

This study helps us understand whether acupuncture is an effective treatment for cyclic mastalgia. By comparing real acupuncture to sham acupuncture, researchers can determine if the improvements seen are due to the acupuncture treatment itself or other factors like the placebo effect.

What does this mean for patients? If you suffer from cyclic mastalgia, this study provides valuable information about the potential benefits of acupuncture as a treatment option. It's important to discuss any treatment options with your health care provider to determine the best approach for your specific situation.

What does this mean for health care providers? This study contributes to the evidence-base for treating cyclic mastalgia with acupuncture. Understanding the results of this study can help health care providers make informed decisions when discussing treatment options with their patients.

Overall, this well-designed study offers insights into the use of acupuncture for cyclic mastalgia, which can be beneficial for both patients and health care providers in making informed decisions about treatment.

DETAILED DESCRIPTION:
A randomized, single-blind, sham acupuncture-controlled trial design was employed, targeting patients with cyclic mastalgia who sought treatment at the Pinggu District Traditional Chinese Medicine Hospital in Beijing, as well as volunteers willing to participate in the trial. Sixty-six patients meeting the inclusion criteria were randomly assigned to two groups: the observation group (acupuncture group) and the control group (sham acupuncture group), with 33 patients in each. The study spanned 16 weeks, divided into two phases: a 4-week baseline period and a 12-week treatment period. The primary outcome measure was the change in daily average overall breast pain assessed using a Visual Analog Scale (VAS). Additionally, infrared temperature changes at the Danzhong (CV17), Rugen (ST18), and Tianzong (SI11) acupoints were observed, and the meridian energy values of the Liver, Spleen, and Stomach meridians were evaluated in the participants.

ELIGIBILITY:
Inclusion Criteria:（1） 18-45 years old; （2）Clinical diagnosis of Cyclic Mastalgia： Breast pain occurs 2 weeks before menstruation, improves after menstruation；（3）The basic rules of menstrual cycle are (28 ± 7) days and 3-7 days （4）Breast X-ray or breast ultrasound examination excludes malignant breast lesions.

Exclusion Criteria:

（1） Received relevant treatment within the past month; （2） with serious cardiovascular and cerebrovascular diseases, severe liver and kidney dysfunction, or coagulation dysfunction; （3）with diseases such as rib cartilage inflammation, chest wall injury, rib fractures, and other external breast pain; （4） in pregnancy or lactation stage; （5）There is a serious skin disease or infection at the intended acupuncture site.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
the change in the daily average Visual Analog Scale (VAS) score for overall breast pain | 1 year
  the change in visual analog scale (VAS) of overall breast pain on a daily basis within the first two weeks before the baseline period and the end of treatment.

SECONDARY OUTCOMES:
the changes in infrared temperature at the acupoints of Danzhong, Rugen, and Tianzong | 1 year
  the changes in infrared temperature at the acupoints of Danzhong, Rugen, and Tianzong
the meridian energy values | 1year
  Evaluate the meridian energy values of the Liver Meridian, Spleen Meridian, and Stomach Meridian in points, with a maximum score of 100 points, using a meridian detector

OTHER OUTCOMES:
effectiveness of the acupuncture blinding | 1 year
  Effectiveness of acupuncture blinding assessed using Jame's BI Index (JBI)，The range of JBI values is 0-1, and the larger the JBI value, the more successful the blind method is.
Treatment-Emergent Adverse Events | 1year
  Safety was determined by recording any adverse reactions or events such as needle sickness, infection, subcutaneous hematoma, subcutaneous nodules, and post-acupuncture pain-including time, severity, treatment measures, and resolution time

IPD SHARING:
Plan to Share IPD: Yes
After the research is completed on December 31, 2026，it will be made available to others upon request to the person in charge (yuchuan106@126.com), only for research, and non-commercial purposes toindividuals affiliated with academic or public health institutions.
Supporting Information: Study Protocol, SAP, CSR
URL: https://register.clinicaltrials.gov/prs/beta/studies/S000F52V00000046/protocol/ipdSharing?edit=true